CLINICAL TRIAL: NCT04055688
Title: Clinical Study of the Utility of a Novel Exoscope System for 5-ALA Fluorescence-Guided Surgery for Gliomas
Brief Title: Novel Exoscope System for 5-ALA Fluorescence-Guided Surgery for Gliomas
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-20014
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Brain Tumor; Glioma
Keywords: Orbeye Surgical Microscope; fluorescence-guided surgery; 5-ALA
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants with known or suspected high grade gliomas
  Interventions: Device: Orbeye surgical videomicroscope; Drug: 5-Aminolevulinic Acid

INTERVENTIONS:
Device: Orbeye surgical videomicroscope — The ORBEYE surgical microscope is an FDA-cleared apparatus designed to facilitate operating procedures that involve fine nerves, blood vessels, and other small anatomic features by providing an enlarged stereoscopic visual field of the surgical site. The 4K 3D digital images of the ORBEYE microscope provide high-resolution stereoscopic images of the fine structures of tissue and blood vessels. As the surgical procedures are displayed on a large 55-inch monitor, the device is expected to reduce fatigue of the operator by eliminating the need for extensive viewing via microscope eyepieces for an extended period of time. The technology adopted in the ORBEYE was developed by Sony Olympus Medical Solutions, and its product design was handled by Olympus Medical Systems Corp. The ORBEYE is marketed by the Olympus Corporation.
Drug: 5-Aminolevulinic Acid — 5- aminolevulinic acid (5-ALA) is a European Medicines Agency- and Food and Drug Administration- (FDA-) approved drug that is administered to patients 2 to 4 hours before surgery and converted preferentially by tumor cells to protoporphyrrin IX (PPIX). PPIX fluoresces red when exposed to blue light. Use of 5-ALA has previously been shown to permit surgeons to obtain a more complete tumor resection, and its use has also been associated with an increased rate of progression-free survival.(3) There are currently 2 surgical microscope systems available on the market that are equipped with a 5-ALA visualization system. These visualization systems are currently classified by the FDA as Class I-exempt accessories to Class I-cleared surgical microscopes.
  Other Names: 5-ALA

SUMMARY:
5-ALA and the Orbeye surgical microscope are U.S. Food and Drug Administration (FDA) approved products. For this study, the Orbeye microscope imaging system is being used with special filters to visualize 5-ALA fluorescence. The FDA currently permits the use of these filters. The purpose of this study is to collect medical information before, during, and after standard treatment in order to better understand how to make this type of procedure accessible to patients.

This study is also being conducted to determine if use of the Orbeye equipped with these special filters improves the ability of the surgeon to remove brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have a suspected or biopsy-proven high-grade glioma (World Health Organization grade II or IV), new or recurrent.
* Indication for craniotomy for removal of a suspected or recurrent brain tumor
* Karnofsky Performance Scale >/- 60%

Exclusion Criteria:

* Prophyria, hypersensitivity to porphyrins
* Renal insufficiency as defined per protocol
* Hepatic insufficiency as defined per protocol
* Existing pregnancy (to be checked by a pregnancy test if of child-bearing age.
* Nursing women or women using inadequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patients at Moffitt Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Compare Visualized Fluroescence within brain tumors | Surgery day one
  6 tissue samples will be obtained intraoperatively for each patient and assessed for 5-ALA visualization (strongly positive.weakly positive/negative). Tissue samples will be submitted for pathological assessment to determine whether tumor cells are present or absent. Visualization results will be evaluated against the pathology results (gold standard) to determine the sensitivity, specificity, positive predictive value and negative predictive value for 5-ALA visualizations with use of the ORBEYE system.

SECONDARY OUTCOMES:
Volume of Residual tumor | up to 48 hours after surgery
  Residual tumor volume will be identified in post surgical MRI scans. Extent of resection will be compared to preoperative MRI scans.
Number of Patients experiencing Adverse Events | Up to 16 days after surgery
  Patients will be assessed for neurological and general side effects/toxicities 7-16 days after surgery.

OTHER OUTCOMES:
Post Surgery Questionnaire | Surgery day one
  Surgeons will complete a questionnaire after each surgery to assess the visual experience of using the ORBEYE during the surgical procedure. The questionnaire asks about the superiority of the ORBEYE system compared to conventional binocular microscope, using a scale of 1-5, 1 being strongly agree and 5 being strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Vogelbaum, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer and Research Institute
Locations (1):
- H. Lee Moffitt Cancer and Research Institute, Tampa, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04055688/ICF_000.pdf